CLINICAL TRIAL: NCT04833439
Title: The Effect of a Fasting MimickINg Diet on the Immune System: an Exploratory Study
Brief Title: The Effect of a Fasting MimickINg Diet on the Immune System
Acronym: FIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.R. Kroep, medical oncologist, associate professor, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL76033.058.21; P21.017 (Other: LUMC)
Record Dates: First submitted 2021-03-30; First posted 2021-04-06 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Healthy Subjects; Cancer; Neoplasms
Keywords: Fasting; Caloric restriction; Immunomodulation; Tumor-Infiltrating Lymphocytes; Fasting Mimicking Diet
MeSH Terms: conditions — Neoplasms; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting Mimicking Diet (Experimental): 2 cycles of 3-day fasting mimicking spaced by a 2 week interval
  Interventions: Other: Fasting Mimicking Diet

INTERVENTIONS:
Other: Fasting Mimicking Diet — Low-caloric, low-protein, plant-based diet regiment for 3 days
  Other Names: Xentigen

SUMMARY:
Fasting or a Fasting Mimicking diet (FMD) can lower blood concentration of glucose and IGF1. Since cancer cells rely mostly on a glucose-based metabolism, FMD renders cancer cells more vulnerable to chemotherapy, thereby enhancing therapeutic efficacy. This process is known as differential stress sensitization (DSS). Another response to nutritional stress by fasting is known as differential stress resistance (DSR). DSR is a state in which healthy cells rather focus resources on protection and internal repair, which can result in reduced chemotherapeutic toxicity. Recent preclinical studies found that fasting or FMD not only aids healthy cell protection, but also has the potential to benefit effector T-cells and could thereby improve antitumor immunity. However in most oncotherapeutic clinical trials investigating the addition of a fasting regimen, other factors such as chemotherapy, surgery and additional medication affect the immune system as well. That is why this explorative study, conducted in healthy subjects, might be more suitable to investigate the immunological alterations upon FMD more specifically. This exploratory study aims to identify immunological alterations by using extensive immunoprofiling before and after three days of FMD in healthy subjects, as well as investigate possible side effects of FMD.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* BMI ≥18.5 and ≤25kg/m2

Exclusion Criteria:

* Chronic disease or active infection
* Medication use other than contraceptive, during the last 12 weeks prior to inclusion.
* A history of allergy
* Blood or plasma donation in the last 12 weeks prior to inclusion.
* Participation in other medical research in the last 12 weeks prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Change in gene expression signature in peripheral blood mononuclear cells (PBMCs) after overnight fast and after completion of 2 cycles of fasting mimicking diet compared to baseline. | 4 weeks
  PBMCs are retrieved from whole blood samples. Gene expression signature is retrieved from PBMCs using RNA-Nanostring technique with the Pancancer IO 360 panel. The Nanostring will report RNA counts for a panel of 770 genes, including 40 housekeeping genes. The data will be normalized on the 40 housekeeping genes for internal control using Nanostring nSolver software. The fold change from baseline to overnight fast and after completion of second fasting mimicking diet will provide insight in affected pathways as well as metabolic and immune signatures.

SECONDARY OUTCOMES:
Change in immune cell properties from PBMCs after overnight fast and after 2 cycles of fasting mimicking diet compared to baseline. | 6 months
  PBMCs retrieved from whole blood samples will be analysed with a 40-plex Aurora flowcytometry panel with markers for T cells and myeloid cells. The flow cytometry will generate frequencies of the different immune cell markers,. A comparison of the frequency data between blood samples will determine change in immune cell properties.
  This analysis will be used to confirm and complement gene expression signature findings on a protein level.
Change in plasma concentration of IGF1, glucose and ketone bodies (Beta-hydroxybutyric acid) after overnight fast and after completion of 2 cycles of fasting mimicking diet compared to baseline. | 4 weeks
  Measured in blood plasma taken at 3 time points.
Percentage of participants reporting adverse events as assessed by CTCAE v5.0 during fasting mimicking diet | 8 weeks
  Descriptive analysis of adverse events by type and grade according to NCI CTCAE v5.0 experienced by participants during fasting mimicking diet assessed after second cycle on day 22.

CONTACTS AND LOCATIONS:
Overall Officials: Judith R Kroep, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No